Data analysis Attention, Teleconferencing and Social Anxiety

Date: 12/05/2022

Identifiers: NCT04729803 Unique Protocol ID: STUDY00000106

## **Data Analysis**

Describe the data analysis plan, including any statistical procedures or power analysis.

## To input text, click in the light grey area below.

We will conduct multi-level models for all analyses (1) to compare the positive and negative interactions, where participants are looking, and social anxiety symptoms; (2) to compare the attention guidance condition to the other exposure groups using the Personal Report of Communication Apprehension as the primary outcome measure. We will use the brms package (Bürkner, 2018) in R to conduct Bayesian multi-level modelling.